CLINICAL TRIAL: NCT04319562
Title: Needle-embedding Therapy Alleviates Depressive Symptoms and Resets the Function of Executive Control System in Subthreshold Depression People: a Randomized Controlled Study
Brief Title: Needle-embedding Therapy Alleviates Depressive Symptoms and Resets the Function of Executive Control System in Subthreshold Depression People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Fu Wenbin, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YN2019ML13
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Subthreshold Depression
Keywords: Subthreshold Depression; Needle-embedding Therapy; Executive Control System

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- needle-embedding therapy (Experimental): The participants in this group will be treated with intradermal thumbtack needle.
  Interventions: Procedure: needle-embedding therapy
- shame needle-embedding therapy (Sham Comparator): The participants in this group will be treated with shame intradermal thumbtack needle.
  Interventions: Device: shame needle-embedding therapy

INTERVENTIONS:
Procedure: needle-embedding therapy — First group is comprised of Xinshu (BL15), Ganshu (BL18), Juque (CV14) bilaterally, and Xin and Gan of auricular point on the left ear. Second group includes Shentang (BL44), Hunmen (BL47), Jiuwei (RN15) bilaterally, and Xin and Gan of auricular point on the right side.
  After skin cleansing with a 75% alcohol swab, intradermal thumbtack needle will be quickly inserted into the skin and embedded at acupoints mentioned above bilaterally. The needles will remain in the acupoints for 3 days and they will be removed by the therapists at next visit. This also can ensure better implementation of the blind method.Participants are required to receive this treatment twice a week. The specification of the needle used in the back shu point is φ9mm 0.20×1.5mm (Seirin® PYONEX; Seirin Corporation, Shizuoka, Japan), that in the auricular point is φ9mm 0.20×0.6mm (Seirin® PYONEX; Seirin Corporation, Shizuoka, Japan).
  Arms: needle-embedding therapy
Device: shame needle-embedding therapy — The acupoint selection in this group is the same as in the needle-embedding therapy group, except that the shame intradermal needles will be used. After skin cleansing with a 75% alcohol swab, the shame intradermal needles，instead of insert into the skin, it can only stick on the surface of the skin. It also will be removed by the therapists after 3 days. This takes place twice a week. The specification of the shame needle is the same as above.
  Arms: shame needle-embedding therapy

SUMMARY:
The main objective of this trial is to evaluate the effectiveness of treating subthreshold depression by needle-embedding therapy. On this basis, the investigators will discuss the mechanism of needle-embedding therapy improving executive function control system.

DETAILED DESCRIPTION:
The needle-embedding therapy is a method of acupuncture, which inserts the intradermal thumbtack needle into skin quickly. The needle will be replaced after 2 or 3 days. This treatment has a great efficacy on subthreshold depression (SD) and it is easy to promote. However, its clinical effect remains to be studied. In this study, the researchers used this method to treat SD by selecting the back shu acupoint and ear acupoint.

This research aims to evaluate the effectiveness of treating subthreshold depression by needle-embedding therapy. On this basis, from the perspective of psychology, this project takes the cognitive function of the SD people as the entry point, in order to find the scientific indicators to quantify the SD people clinically from the perspective of the executive function control system. At the same time, magnetic resonance imaging(MRI) was used to compare and analyze the brain executive control system of subthreshold depression group and normal group, and to observe the specificity of brain structure, network and function of subthreshold depression group. Finally, through the comparative analysis of the brain executive control system of the subthreshold depression group with intradermal thumbtack needle therapy and shame intradermal thumbtack needle therapy, the neural mechanism of needle-embedding therapy promoting the function reset of the brain executive control system was speculated based on the evaluation of the efficacy of needle-embedding therapy.

80 patients will be divided into two groups randomly, intradermal thumbtack needle group or shame intradermal thumbtack needle group, and evaluated before and after intervention.

The primary study outcomes will be depressive symptoms as measured by the PHQ-9. Secondary outcomes will be the ability of executive control system, health-related quality of life and anxiety symptoms measured as described previously. Tertiary outcomes will be the difference between the results of fMRI of SD people and normal brain database, and the difference between the treatment group and control group, which can observe the specificity of brain structure, network and function in subthreshold depression.

The results will be analyzed and presented descriptively, as of statistical comparisons of pre- and post-treatment and the relationship between the groups.

ELIGIBILITY:
Inclusion Criteria:

Applicants self-identifying with a diminished mood who

* screened positive for subthreshold depressive symptoms (Centre for Epidemiological Studies Depression Scale (CES-D) ≥ 16;
* were scheduled for a semistructural clinical interview (the Mini International Neuropsychiatric Interview, the MINI) conducted by specialists in psychiatry to diagnose whether they are SD；
* were not currently receiving or had a plan to receive a psychotherapy for any kind of mental health problem；
* had had no psychotherapy for any kind of mental health disorder in the past six months.

Exclusion Criteria:

patients had

* antidepressant use
* alcohol dependency
* psychosis
* recent suicidalrisk
* significant cognitive impairment
* recent bereavement
* terminal illness on clinical grounds

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms as assessed by Patient Health Questionnaire-9（PHQ-9） | Baseline and 6 weeks, 1-, 3-, 6- and 12-month follow-up
  The PHQ-9 questionnaire can directly reflect the subjective feelings of depressed patients and their changes in treatment. As a severity measure, the PHQ-9 score can range from 0 to 27. since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). The higher the score, the more severe the depressive symptoms.

SECONDARY OUTCOMES:
Change of attention network test(ANT) | Baseline and 6 weeks
  Combined with spatial cue task and flanker task, Attention Network Test can effectively measure different Attention Network effects. ANT can represent three different attention networks (alertness effect, orientation effect and executive control effect).
Change of psychomotor vigilance task (PVT) | Baseline and 6 weeks
  The psychomotor vigilance task (PVT) is a sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus. Research indicates increased sleep debt or sleep deficit correlates with deteriorated alertness, slower problem-solving, declined psycho-motor skills, and increased rate of false responding.
Change in health-related quality of life as assessed by Short Form Survey (SF-12). | Baseline and 6 weeks, 1-, 3-, 6- and 12-month follow-up
  This questionnaire can reflect the patients' health-related quality of life.SF-12 score ranges from 0 [lowest level of health] to 100 [highest level of health].
Change in anxiety symptoms as assessed by Generalized Anxiety Disorder Assessment (GAD-7). | Baseline and 6 weeks, 1-, 3-, 6- and 12-month follow-up
  This questionnaire can reflect the anxiety symptoms of patients.GAD-7 score ranges from 0 [no anxiety] to 21 [severe anxiety].

OTHER OUTCOMES:
Difference of Functional magnetic resonance imaging scans between two group. | Baseline and 6 weeks
  Before the intervention, 40 people were randomly selected to complete the fMRI examination, and the results were compared with the normal brain database. After the intervention, all subjects underwent MR examination, and the treatment group and the control group were compared with each other.
  The signal of the function, gray matter fiber and white matter fiber of the dorsolateral prefrontal cortex (DLPFC) were extracted from the resting-state fMRI data. These signal will be calculated the functional network of the brain based on graph theory. Therefore, the investigator will compare the difference between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Webin Fu, MD, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- The Second Affiliated hospital of Guangzhou University of Chinese Medicine (Guangdong Provincial Hospital of Chinese Medicine), Guangzhou, Guangdong, China